CLINICAL TRIAL: NCT06623279
Title: A Phase 1, Open-label, Multiple-cohort, Dose-escalation Study to Evaluate the Safety and Tolerability of HG202 High-fidelity CRISPR-Cas13 (hfCas13Y) RNA-targeting Therapy for Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: Open-laBel Dose-escalation Study for CRISPR/cas13- Rna TargetInG THerapy for the Treatment of Neovascular Age-related Macular Degeneration in Phase I Trial
Acronym: BRIGHT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HuidaGene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HG20202
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD)
Keywords: Macular Degeneration; nAMD; wAMD; Gene-editing; CRISPR; HG202
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Three dosing cohort:
  Low dose : 3 subjects Middle dose: 6 subjects High dose: 6 subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HG202 (Experimental): The study will enroll up to 3 dose cohorts：Low dose/Middle dose/High dose
  Interventions: Genetic: HG202

INTERVENTIONS:
Genetic: HG202 — Method of Administration: Once unilateral subretinal injection; The duration of the study includes a 4-week screening period, enrollment visit, treatment visit and 52 weeks follow-up period, 4 more years long term follow up as an extension study.

SUMMARY:
Age-related macular degeneration (AMD) leads to severe and irreversible vision loss, while neovascular AMD (nAMD) accounts for 80-90% of AMD blindness. Current anti-VEGF therapies are the standard of care, but these therapies require life-long repeated intraocular injections. These frequent intravitreal injections increase the risk of complications, including submacular hemorrhage, intraocular hypertension, inflammation, and retinal detachment. Therefore, repeated treatments for nAMD place a substantial burden on healthcare systems, patients, and their caregivers. Additionally, approximately 25-35% of individuals with aggressive nAMD show suboptimal responses to the anti-VEGF therapies, experience treatment-extended failure, or require intensive, frequent intraocular injections, and do not prevent irreversible vision loss.

HG202 is a CRISPR/Cas13 RNA-editing therapy delivered through one single AAV vector to partially knock down the expression of VEGFA and thus inhibit CNV formation in AMD. The long-term, stable delivery of HG202 following a one-time gene-editing therapy treatment for nAMD may potentially reduce the frequent injections and the potential risks of currently available anti-VEGF therapies since it does not rely on the long-term expression of anti-VEGF antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 50 and ≤ 85 years at the time of signing the ICF;
* Active macular choroidal neovascularization (MNV) secondary to nAMD in the study eye;
* Sentinel (1st) subject for each dose cohort must have a BCVA ≤ 20/63 and ≥ 20/400 (≤63 and ≥ 19 ETDRS letters) in the study eye. Following the sentinel subject evaluation, the rest of the subjects in the dose cohort must have a BCVA between ≤ 20/40 and ≥ 20/400 (≤ 73 and ≥ 19 ETDRS letters) in the study eye.
* Able to perform visual acuity and retinal function tests and able and willing to comply with study procedures for this clinical trial.

Exclusion Criteria:

* Retinal or subretinal hemorrhage, scarring, or fibrosis of greater than 50% of the total lesion in the study eye;
* Other ocular diseases that may affect central vision in the study eye;
* Any other cause of CNV than nAMD in the study eye
* Uncontrolled glaucoma in the study eye;
* History or presence of corneal transplant or corneal dystrophy in the study eye;
* History of other intraocular surgery in the study eye within 3 months prior to baseline;
* Prior gene therapy or oligonucleotide therapy;
* Other conditions judged by the investigator as inappropriate for the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular and systemic adverse events | 52 weeks
  Number of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Mean change from baseline in best-corrected visual acuity (BCVA) | 52 weeks
  Change from baseline in BCVA as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) chart in the study eye at different doses
Mean change in annualized rate of supplemental injections | 52 weeks
  Change from baseline in the number of anti-VEGF injections which is annualized to a per year rate in the study eye at different doses

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — HuidaGene Therapeutics Co., Ltd.